CLINICAL TRIAL: NCT06547515
Title: Bone and Muscle Health Following Sleeve Gastrectomy in Men, Premenopausal and Postmenopausal Women
Acronym: BONUS
Status: Recruiting | Type: Observational
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Claudia Gagnon, Principal Investigator, Endocrinologist, Regular Researcher of the Endocrinology-Nephrology Axis, CHU de Quebec-Universite Laval
Other Study IDs: MP-10-2022-3823
Record Dates: First submitted 2024-07-25; First posted 2024-08-09 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Bariatric Surgery; Bone Health; Severe Obesity; Muscle Health
Keywords: bariatric surgery; Bone health; Severe Obesity; Muscle Health
MeSH Terms: conditions — Obesity, Morbid | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Biospecimen Retention: Samples With DNA — Blood (serum and plasma)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Sleeve gastrectomy - Men: n = 39 men with obesity undergoing sleeve gastrectomy
  Interventions: Procedure: Bariatric surgery
- Sleeve gastrectomy - Premenopausal women: n = 39 premenopausal women with obesity undergoing sleeve gastrectomy
  Interventions: Procedure: Bariatric surgery
- Sleeve gastrectomy - Postmenopausal women: n = 39 postmenopausal women with obesity undergoing sleeve gastrectomy
  Interventions: Procedure: Bariatric surgery
- Obese non-surgical group: n = 39 (13 men, 13 premenopausal and 13 postmenopausal women) obese non-surgical individuals

INTERVENTIONS:
Procedure: Bariatric surgery — Sleeve gastrectomy
  Groups: Sleeve gastrectomy - Men; Sleeve gastrectomy - Postmenopausal women; Sleeve gastrectomy - Premenopausal women

SUMMARY:
Background: Bariatric surgery is gaining in popularity. While it's health benefits are undisputed, the older malabsorptive bariatric procedures (Roux-in-Y gastric bypass - RYGB and biliopancreatic diversion - BPD) are associated with an increased risk of fractures and falls as early as 3-5 years after surgery. Sleeve gastrectomy - SG is now the most performed bariatric procedure. Although SG does not cause malabsorption, it is predicted to result in bone and muscle loss via weight loss and weight loss-independent mechanisms. Primary aim: to compare the changes in spine volumetric bone mineral density (vBMD) by quantitative computed tomography (QCT) and muscle mass at mid-femur by computed tomography (CT) at 3 years in the 3 groups of: 1) men; 2) premenopausal women; 3) postmenopausal women after SG versus their respective non-surgical peers who did not undergo SG in the 3-year period following recruitment. Secondary aims: to compare the changes in vBMD by QCT at skeletal sites other than the spine and in areal bone mineral density (aBMD) by dual-energy X-ray absorptiometry (DXA), whole-body muscle mass by DXA, muscle quality by CT at mid-femur and muscle strength as well as in selected physical performance and capacity tests shown to predict falls and fractures between 0-1 and 1-3 years after SG in the same 3 groups after SG vs. in the respective non-surgical groups.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged >18 years;
* Awaiting SG for the bariatric group or meeting the criteria for SG but not undergoing surgery for the non-surgical group.
* Menopause: defined as the absence of menses for a year and a serum follicular-stimulating hormone (FSH) >40 UI/L.
* Women taking oral contraceptive pills or hormone replacement therapy
* Patients with type 2 diabetes.

Exclusion Criteria:

* Type 1 diabetes;
* Disease (e.g., uncontrolled thyroid disease, Malabsorptive or overt inflammatory disorder)
* Metabolic bone disease other than osteoporosis or type 2 diabetes,
* Creatinine clearance <30 ml/min) or medication (e.g., glucocorticoids, anti-epileptic drugs, osteoporosis therapy, thiazolidinediones) affecting bone metabolism;
* Weight >204 kg (DXA weight limit) or BMI >60 kg/m2 (upper limit to allow for QCT examination);
* Current or planned pregnancy during follow-up; breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Gender role has been shown to influence lifestyle behaviours such as physical activity and nutrition. It is however unknown whether gender role influences adherence to the American Society for Metabolic and Bariatric Surgery physical activity and dietary intake/supplement recommendations that are important for bone/muscle health after bariatric surgery. A short questionnaire, the validated 12-item Bem Sex Role Inventory, will be administered to the participants to categorize them into 4 gender role categories. In an exploratory descriptive analysis, the investigators will calculate the proportion of participants in each gender role category meeting the dietary/supplement intake and physical activity recommendations and document the type and amount of physical activity they perform.
Study Population: This is a multicentre, prospective and observational study comprising a SG bariatric group undergoing SG (n=117) comprising an equal number of men, premenopausal and postmenopausal women (n=39/group) meeting the inclusion/exclusion criteria, and assessed before, and at one and 3 years after SG. An obese non-surgical group (n=39; 13 men, premenopausal and postmenopausal women) meeting the criteria for SG but who will not undergo surgery during the 3-year period following recruitment will be assessed using the same tests and at the same timepoints.
Sampling Method: Probability Sample
Enrollment: 156 (Estimated)
Dates: Start 2022-09-14 (Actual); Primary Completion 2026-08-15 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
Change in vBMD at the spine (L2-L3) and proximal femur | before, 1 year after and 3 years after bariatric surgery
  assessed by QCT
Change in muscle mass at mid-femur | before, 1 year after and 3 years after bariatric surgery
  determined by measuring cross-sectional area at mid-femur (CT)

SECONDARY OUTCOMES:
Change in vBMD at skeletal sites other than the spine | before, 1 year after and 3 years after bariatric surgery
  assessed by QCT
Change in aBMD at skeletal sites | before, 1 year after and 3 years after bariatric surgery
  assessed by DXA
Change in whole body muscle mass | before, 1 year after and 3 years after bariatric surgery
  assessed by DXA
Change in muscle quality at mid-femur | before, 1 year after and 3 years after bariatric surgery
  muscle fat infiltration, using CT attenuation in Hounsfield unit (HU)
Change in muscle strength | before, 1 year after and 3 years after bariatric surgery
  assessed by CT
Change in upper extremity muscle strength | before, 1 year after and 3 years after bariatric surgery
  by hand grip strength
Change in lower extremity muscle strength | before, 1 year after and 3 years after bariatric surgery
  knee extensor strength
Change in muscle mass (muscle cross-sectional area) and function | before, 1 year after and 3 years after bariatric surgery
  by timed up and go test
Change in muscle mass (muscle cross-sectional area) and function | before, 1 year after and 3 years after bariatric surgery
  by 6-minute walk test

OTHER OUTCOMES:
The clinical impact of SG on self-reported falls | before, 1 year after and 3 years after bariatric surgery
  by self-reported questionnaire (yes/No)
The clinical impact of SG on self-reported incidence of vertebral and non-vertebral fractures | before, 1 year after and 3 years after bariatric surgery
  by questionnaire (yes/No and number of fractures, how)
The proportion of participants meeting the recommendations for physical activity | before, 1 year after and 3 years after bariatric surgery
  by international physical activity questionnaire short version (score in MET-min/week), (Min 495 MET-minute/week, Max 1200 MET-minute/week)
The proportion of participants meeting the recommendations for dietary protein intake | before, 1 year after and 3 years after bariatric surgery
  Dietary journal, Calculating macronutrient and micronutrient intake per day 3 web-based 24-h recalls
The proportion of participants meeting the recommendations for calcium and vitamin D intake from diet and supplements | before, 1 year after and 3 years after bariatric surgery
  serum D vitamin (25ODH) in blood sample
The proportion of participants meeting the recommendations for calcium and vitamin D intake from diet and supplements | before, 1 year after and 3 years after bariatric surgery
  Parathyroid hormone (PTH) in blood sample
Changes in C-Telopeptide, amino-terminal propeptide of type 1 procollagen (P1NP), osteocalcin | before, 1 year after and 3 years after bariatric surgery
  assessed by blood sample. unit: micro g/l
Changes in calcium, | before, 1 year after and 3 years after bariatric surgery
  assessed by blood sample. unit: mmol/l
Changes in albumin, | before, 1 year after and 3 years after bariatric surgery
  assessed by blood sample. unit:g/l
Changes in creatinin | before, 1 year after and 3 years after bariatric surgery
  assessed by blood sample. unit: micromol/l
Changes in folliculo-stimulant (FSH) | FSH will be measured at the time of surgery, when women had withdrawn their hormones for 3 months preceding surgery.
  assessed by blood sample. unit: UI/l
  FSH will help categorize hysterectomized women or those with non-menopausal amenorrhea. Premenopause will be defined as menses in the last year.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Gagnon, Dr, Principal Investigator — CHU de Québec - Université Laval
Locations (1):
- Centre de recherche de l'IUCPQ, Québec, Canada